CLINICAL TRIAL: NCT02883686
Title: The Effectiveness of the Alma Peer Mentoring Program for Pregnant Women With Depression
Brief Title: Randomized Controlled Trial of the Alma Peer Mentoring Program for Pregnant Women Experiencing Depression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Kaiser Permanente (Other); Emory University (Other)
Responsible Party: Principal Investigator, Sona Dimidjian, Professor, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO-16-2391
Record Dates: First submitted 2016-08-03; First posted 2016-08-30 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Depression; Depression, Postpartum
Keywords: Perinatal Depression; Postpartum Depression; Pregnancy; Peer-delivered; Task-sharing
MeSH Terms: conditions — Depression; Depression, Postpartum | interventions — N(alpha)-acetyllysine-N-methylamide

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to the Alma intervention or to Usual Care
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alma Mentoring plus usual care (Experimental): Alma peer-mentoring
  Interventions: Behavioral: Alma
- Enhanced Usual Care (No Intervention): Usual care for depression within the Kaiser Permanente of Colorado healthcare system plus study monitoring of depression symptoms and feedback.

INTERVENTIONS:
Behavioral: Alma — Alma peer-mentoring
  Arms: Alma Mentoring plus usual care

SUMMARY:
Women have double the odds of getting depressed as men and commonly experience depression during the childbearing and early parenting years. Many new and expectant mothers who experience depression never receive help. Alma is a new program, collaboratively developed by a team of researchers, clinicians, and mothers who have personal experience with depression, to support women experiencing depression during pregnancy and the postpartum period. In the Alma program, mothers who themselves have experienced and recovered from depression during the perinatal period, are trained to provide peer mentoring to depressed new and expectant mothers. Peer mentors are trained by professionals who are experts in using skills to recover from depression. These skills are informed by an evidence-based framework called Behavioral Activation (BA). Peer mentors do not provide psychotherapy and are not licensed mental health providers.

DETAILED DESCRIPTION:
Women have double the odds of getting depressed as men and commonly experience depression during the childbearing and early parenting years. Many new and expectant mothers who experience depression never receive help.

Alma is a new program, collaboratively developed by a team of researchers, clinicians, and mothers who have personal experience with depression, to support women experiencing depression during pregnancy and the postpartum period. We call this program Alma because the meaning of the word, in English and Spanish, captures what we hope moms will feel when they connect with this program. In English, the meaning comes from the Latin word for "nourishing" and "kind," and in Spanish, the meaning is "soul." Through the unique synergy of science and community, the Alma program provides the tools and support needed to nourish moms in supporting their own well-being.

In the Alma program, mothers who themselves have experienced and recovered from depression during the perinatal period, are trained to provide peer mentoring to depressed new and expectant mothers. Peer mentors are trained to provide 6-10 mentoring meetings with each of the new and expectant mothers with whom they are paired. The peer mentors are trained by professionals who are experts in using skills to recover from depression. These skills are informed by an evidence-based framework called Behavioral Activation (BA). Peer Mentors are trained to support and encourage self-monitoring, scheduling activities, solving problems, and bridging to informal and formal professional support. Peer mentors draw on their training and own lived experience to provide hope and reduce the social isolation and stigma associated with perinatal depression. Among the evidence-based approaches to help people recover from depression, Alma uses BA as a lens because many studies have demonstrated that these skills are effective in recovering from depression. It has been provided in a self-guided format and by lay counselors and licensed mental health providers. Peer mentors do not provide psychotherapy and are not licensed mental health providers.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled member of Kaiser Permanente of Colorado (KPCO)
* Current PHQ-9 score greater than or equal to 10
* Current Columbia-Suicide Severity Rating Scale (C-SSRS) score less than 3
* Currently pregnant

Exclusion Criteria:

* Lifetime diagnosis of bipolar disorder or psychotic symptoms
* Dementia or cognitive impairment disorder recorded in the medical record
* Current substance abuse behavior
* At immediate risk of self-harm
* Unable to speak and read English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2020-04-28 (Actual); Study Completion 2020-04-28 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire (PHQ-9) score | Every 2 weeks for the first 12 weeks of the study, then monthly until 3-months postpartum
  Self-report measure of depression symptoms.

SECONDARY OUTCOMES:
Change in Generalized Anxiety Disorder Questionnaire (GAD-7) score | Every 2 weeks for the first 12 weeks of the study, then monthly until 3-months postpartum
  Self-report measure of generalized anxiety symptoms.
Change in Perceived Stress Scale (PSS-10) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report measure of stress.
Change in WHO Disability Assessment Schedule (WHODAS 2.0) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report measure of health, disability, and functioning.
Parenting Stress Index-Short Form (PSI-4/SF) | 3-months postpartum
  Self-reported stress in the parent-child system.
Change in Behavioral Activation for Depression Scale (BADS) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report questionnaire that assesses activation in daily life: Activation, Avoidance/Rumination, Work/School Impairment, and Social Impairment.
Change in Reward-Probability Index (RPI) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report questionnaire that assess proxy dimensions of response-contingent positive reinforcement: reward probability and environmental suppressors inhibiting access to reinforcement.
Change in Environmental Reward Observation Scale (EROS) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report questionnaire that assess the experience of environmental reward over the past several weeks.
Change in Attitudes Toward Motherhood (AToM) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report questionnaire that assess women's attitudes about motherhood, including beliefs related to others' judgments, beliefs about maternal responsibility, and maternal role idealization.
Working Alliance Inventory - Short Form (Intervention group only) | 12-weeks post-randomization
  Self-report questionnaire that assess participant's working alliance with their peer mentor.
Change in Self- Compassion Scale (SCS) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report measure of self-compassion.
Mother Inventory of Reward Experiences (MIRE) | 3-months postpartum
  Self-report questionnaire assessing reward responsivity in parenting.
Change in Social Support Questionnaire - Short Form (SSQ-SF) score | Baseline, 12-weeks post-randomization, 3-months postpartum
  Self-report questionnaire assessing social support available to a participant and their perception of the quality of that social support.
Client Satisfaction Questionnaire (CSQ-8) | 12-weeks post-randomization
  Self-report measure of general satisfaction with the Alma program. Participants randomized to treatment as usual will receive a CSQ-8 to measure general satisfaction with Kaiser Permanente of Colorado mental health services.
Change in Effort-Expenditure for Rewards Task (EEfRT) performance | Baseline, 12-weeks post-randomization, 3-months postpartum
  Computerized behavior task administered remotely that assesses effort-based decision-making.
Change in Experience Sampling Survey response | Baseline, 12-weeks post-randomization, 3-months postpartum
  Momentary mood and activity assessed by self-report triggered by text-message prompt to complete a survey.
Change in Go/No-Go Task (GNAT) performance | Baseline, 12-weeks post-randomization, 3-months postpartum
  Computerized behavior task administered remotely that assesses implicit associations pairing the self with both stigma and belonging.
Exit Interview | 3-months postpartum
  An Exit Interview will be administered to solicit participant feedback about the Alma program and recommendations for improvement, including questions about overall program and specific Alma components, including telephone- or videoconference- based delivery, length and number of sessions, spacing between sessions, peer characteristics, and ease of access to peers.

CONTACTS AND LOCATIONS:
Overall Officials: Sona Dimidjian, PhD, Principal Investigator — University of Colorado, Boulder; Arne Beck, PhD, Principal Investigator — Kaiser Permanente
Locations (2):
- United States (2):
  - Kaiser Permanente of Colorado, Aurora, Colorado
  - University of Colorado Boulder, Boulder, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study information website for potential participants. — http://almastudy.kp.org/